CLINICAL TRIAL: NCT03581032
Title: Optimization of Cardiac Pacing Using CardioMEMS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St. Francis Hospital, New York (Other)
Responsible Party: Principal Investigator, Rita Jermyn, MD, Director of Center for Cardiac Therapeutics, St. Francis Hospital, New York
Other Study IDs: 17-13
Record Dates: First submitted 2018-05-25; First posted 2018-07-10 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A-Active reprogram follwed by sham: This arm will be randomized to have PACING device reprogramming followed by sham reprogramming
  Interventions: Device: Active reprogam
- B-Sham followed by active reprogram: This arm will be randomized to have sham reprogramming followed by active pacing reprogramming
  Interventions: Device: Active reprogam

INTERVENTIONS:
Device: Active reprogam — Reprogram Changes in AV/PV delays

SUMMARY:
This study is designed to determine if a simplified technique for cardiac device reprogramming using pulmonary artery pressure (PAP) data in the acute setting holds promise to improve subjective assessments of patient quality of life (QOL), objective measurements of functional capacity, and specific systolic and diastolic echocardiographic indices.

DETAILED DESCRIPTION:
The present study is designed to determine if a simplified technique for cardiac device( CRT) reprogramming using pulmonary artery pressure (PAP) via implanted CardioMEMS device data in the acute setting holds promise to improve subjective assessments of patient quality of life (QOL), objective measurements of functional capacity, and specific systolic and diastolic echocardiographic indices. The protocol requires prospective collection and analysis of echocardiographic data, subjective symptoms (Minnesota Living with Heart Failure Questionnaires), and 6-minute walk distance measurements in patients with implanted biventricular pacemakers / defibrillators who are predominantly ventricularly paced, in normal sinus rhythm, have documented NYHA class 3 Heart Failure, and have implanted pulmonary artery pressure monitors (CardioMEMS, St. Jude Medical CRMD, St. Paul, MN). Data collection will occur at presentation (rest and with ambulation), one month post-reprogramming, and two months after evaluation and / or reprogramming.

ELIGIBILITY:
Inclusion Criteria:

1. Patients have implanted PPM, ICD, or CRT devices and CardioMEMS
2. Patients can ambulate for 6 minutes and lay on a flat surface
3. Patients are paced > 95% of the time
4. Patients are not in acute CHF and are on a stable medication regimen
5. Patients have adequate echocardiographic windows
6. Patients can consent independently

Exclusion Criteria:

1. Patients with poor echocardiographic acoustical resolution.
2. Patients with congenital heart disease.
3. Patients with mechanical aortic or mitral valve replacements.
4. Patients with significant mitral annular calcification.
5. Patients with irregular heart rates: atrial fibrillation, supraventricular tachycardia, atrial premature contractions, and ventricular arrhythmia that would preclude data acquisition.
6. Patients unable to remain still secondary to movement disorders or agitation.
7. Inpatient status
8. Patients with poorly controlled HTN (SBP>160/90

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Subject Recruitment Subjects will be recruited from the CHF outpatient clinic at St Francis Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Pulmonary artery pressure changes | 30 days
  Primary endpoint is changes in of pulmonary artery pressures within 30 days in patients who have optimization of pacing devices.

CONTACTS AND LOCATIONS:
Overall Officials: Rita Jermyn, MD, Principal Investigator — Saint Francis Hospital
Locations (1):
- St Francis Hospital, Roslyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abraham WT, Fisher WG, Smith AL, Delurgio DB, Leon AR, Loh E, Kocovic DZ, Packer M, Clavell AL, Hayes DL, Ellestad M, Trupp RJ, Underwood J, Pickering F, Truex C, McAtee P, Messenger J; MIRACLE Study Group. Multicenter InSync Randomized Clinical Evaluation. Cardiac resynchronization in chronic heart failure. N Engl J Med. 2002 Jun 13;346(24):1845-53. doi: 10.1056/NEJMoa013168. PMID 12063368
- [Result] Young JB, Abraham WT, Smith AL, Leon AR, Lieberman R, Wilkoff B, Canby RC, Schroeder JS, Liem LB, Hall S, Wheelan K; Multicenter InSync ICD Randomized Clinical Evaluation (MIRACLE ICD) Trial Investigators. Combined cardiac resynchronization and implantable cardioversion defibrillation in advanced chronic heart failure: the MIRACLE ICD Trial. JAMA. 2003 May 28;289(20):2685-94. doi: 10.1001/jama.289.20.2685. PMID 12771115
- [Result] Chung ES, Leon AR, Tavazzi L, Sun JP, Nihoyannopoulos P, Merlino J, Abraham WT, Ghio S, Leclercq C, Bax JJ, Yu CM, Gorcsan J 3rd, St John Sutton M, De Sutter J, Murillo J. Results of the Predictors of Response to CRT (PROSPECT) trial. Circulation. 2008 May 20;117(20):2608-16. doi: 10.1161/CIRCULATIONAHA.107.743120. Epub 2008 May 5. PMID 18458170
- [Result] Mullens W, Grimm RA, Verga T, Dresing T, Starling RC, Wilkoff BL, Tang WH. Insights from a cardiac resynchronization optimization clinic as part of a heart failure disease management program. J Am Coll Cardiol. 2009 Mar 3;53(9):765-73. doi: 10.1016/j.jacc.2008.11.024. PMID 19245967
- [Result] Birnie D, Lemke B, Aonuma K, Krum H, Lee KL, Gasparini M, Starling RC, Milasinovic G, Gorcsan J 3rd, Houmsse M, Abeyratne A, Sambelashvili A, Martin DO. Clinical outcomes with synchronized left ventricular pacing: analysis of the adaptive CRT trial. Heart Rhythm. 2013 Sep;10(9):1368-74. doi: 10.1016/j.hrthm.2013.07.007. Epub 2013 Jul 11. PMID 23851059
- [Result] Martin DO, Lemke B, Birnie D, Krum H, Lee KL, Aonuma K, Gasparini M, Starling RC, Milasinovic G, Rogers T, Sambelashvili A, Gorcsan J 3rd, Houmsse M; Adaptive CRT Study Investigators. Investigation of a novel algorithm for synchronized left-ventricular pacing and ambulatory optimization of cardiac resynchronization therapy: results of the adaptive CRT trial. Heart Rhythm. 2012 Nov;9(11):1807-14. doi: 10.1016/j.hrthm.2012.07.009. Epub 2012 Jul 14. PMID 22796472
- [Result] Starling RC, Krum H, Bril S, Tsintzos SI, Rogers T, Hudnall JH, Martin DO. Impact of a Novel Adaptive Optimization Algorithm on 30-Day Readmissions: Evidence From the Adaptive CRT Trial. JACC Heart Fail. 2015 Jul;3(7):565-572. doi: 10.1016/j.jchf.2015.03.001. Epub 2015 Jun 10. PMID 26071616
- [Result] Galderisi M, Benjamin EJ, Evans JC, D'Agostino RB, Fuller DL, Lehman B, Wolf PA, Levy D. Intra- and interobserver reproducibility of Doppler-assessed indexes of left ventricular diastolic function in a population-based study (the Framingham Heart Study). Am J Cardiol. 1992 Nov 15;70(15):1341-6. doi: 10.1016/0002-9149(92)90772-q. PMID 1442588
- [Result] Ritter P, Padeletti L, Gillio-Meina L, Gaggini G. Determination of the optimal atrioventricular delay in DDD pacing. Comparison between echo and peak endocardial acceleration measurements. Europace. 1999 Apr;1(2):126-30. doi: 10.1053/eupc.1998.0032. PMID 11228855
- [Result] Meluzin J, Novak M, Mullerova J, Krejci J, Hude P, Eisenberger M, Dusek L, Dvorak I, Spinarova L. A fast and simple echocardiographic method of determination of the optimal atrioventricular delay in patients after biventricular stimulation. Pacing Clin Electrophysiol. 2004 Jan;27(1):58-64. doi: 10.1111/j.1540-8159.2004.00386.x. PMID 14720156
- [Result] Kindermann M, Frohlig G, Doerr T, Schieffer H. Optimizing the AV delay in DDD pacemaker patients with high degree AV block: mitral valve Doppler versus impedance cardiography. Pacing Clin Electrophysiol. 1997 Oct;20(10 Pt 1):2453-62. doi: 10.1111/j.1540-8159.1997.tb06085.x. PMID 9358487
- [Result] Sawhney NS, Waggoner AD, Garhwal S, Chawla MK, Osborn J, Faddis MN. Randomized prospective trial of atrioventricular delay programming for cardiac resynchronization therapy. Heart Rhythm. 2004 Nov;1(5):562-7. doi: 10.1016/j.hrthm.2004.07.006. PMID 15851220
- [Result] Butter C, Stellbrink C, Belalcazar A, Villalta D, Schlegl M, Sinha A, Cuesta F, Reister C. Cardiac resynchronization therapy optimization by finger plethysmography. Heart Rhythm. 2004 Nov;1(5):568-75. doi: 10.1016/j.hrthm.2004.07.002. PMID 15851221
- [Result] Perego GB, Chianca R, Facchini M, Frattola A, Balla E, Zucchi S, Cavaglia S, Vicini I, Negretto M, Osculati G. Simultaneous vs. sequential biventricular pacing in dilated cardiomyopathy: an acute hemodynamic study. Eur J Heart Fail. 2003 Jun;5(3):305-13. doi: 10.1016/s1388-9842(02)00204-0. PMID 12798828
- [Result] van Gelder BM, Bracke FA, Meijer A, Lakerveld LJ, Pijls NH. Effect of optimizing the VV interval on left ventricular contractility in cardiac resynchronization therapy. Am J Cardiol. 2004 Jun 15;93(12):1500-3. doi: 10.1016/j.amjcard.2004.02.061. PMID 15194020
- [Result] Yu CM, Fung JW, Zhang Q, Chan CK, Chan YS, Lin H, Kum LC, Kong SL, Zhang Y, Sanderson JE. Tissue Doppler imaging is superior to strain rate imaging and postsystolic shortening on the prediction of reverse remodeling in both ischemic and nonischemic heart failure after cardiac resynchronization therapy. Circulation. 2004 Jul 6;110(1):66-73. doi: 10.1161/01.CIR.0000133276.45198.A5. Epub 2004 Jun 14. PMID 15197148
- [Result] Lee KL, Burnes JE, Mullen TJ, Hettrick DA, Tse HF, Lau CP. Avoidance of right ventricular pacing in cardiac resynchronization therapy improves right ventricular hemodynamics in heart failure patients. J Cardiovasc Electrophysiol. 2007 May;18(5):497-504. doi: 10.1111/j.1540-8167.2007.00788.x. Epub 2007 Apr 11. PMID 17428272
- [Result] van Gelder BM, Bracke FA, Meijer A, Pijls NH. The hemodynamic effect of intrinsic conduction during left ventricular pacing as compared to biventricular pacing. J Am Coll Cardiol. 2005 Dec 20;46(12):2305-10. doi: 10.1016/j.jacc.2005.02.098. PMID 16360063
- [Result] Thibault B, Ducharme A, Harel F, White M, O'Meara E, Guertin MC, Lavoie J, Frasure-Smith N, Dubuc M, Guerra P, Macle L, Rivard L, Roy D, Talajic M, Khairy P; Evaluation of Resynchronization Therapy for Heart Failure (GREATER-EARTH) Investigators. Left ventricular versus simultaneous biventricular pacing in patients with heart failure and a QRS complex >/=120 milliseconds. Circulation. 2011 Dec 20;124(25):2874-81. doi: 10.1161/CIRCULATIONAHA.111.032904. Epub 2011 Nov 21. PMID 22104549
- [Result] Yu CM, Wang L, Chau E, Chan RH, Kong SL, Tang MO, Christensen J, Stadler RW, Lau CP. Intrathoracic impedance monitoring in patients with heart failure: correlation with fluid status and feasibility of early warning preceding hospitalization. Circulation. 2005 Aug 9;112(6):841-8. doi: 10.1161/CIRCULATIONAHA.104.492207. Epub 2005 Aug 1. PMID 16061743
- [Result] Khoury DS, Naware M, Siou J, Blomqvist A, Mathuria NS, Wang J, Shih HT, Nagueh SF, Panescu D. Ambulatory monitoring of congestive heart failure by multiple bioelectric impedance vectors. J Am Coll Cardiol. 2009 Mar 24;53(12):1075-81. doi: 10.1016/j.jacc.2008.12.018. PMID 19298923
- [Result] Maines M, Catanzariti D, Cemin C, Vaccarini C, Vergara G. Usefulness of intrathoracic fluids accumulation monitoring with an implantable biventricular defibrillator in reducing hospitalizations in patients with heart failure: a case-control study. J Interv Card Electrophysiol. 2007 Sep;19(3):201-7. doi: 10.1007/s10840-007-9155-4. Epub 2007 Sep 6. PMID 17805952
- [Result] Small RS, Wickemeyer W, Germany R, Hoppe B, Andrulli J, Brady PA, Labeau M, Koehler J, Sarkar S, Hettrick DA, Tang WH. Changes in intrathoracic impedance are associated with subsequent risk of hospitalizations for acute decompensated heart failure: clinical utility of implanted device monitoring without a patient alert. J Card Fail. 2009 Aug;15(6):475-81. doi: 10.1016/j.cardfail.2009.01.012. Epub 2009 Mar 17. PMID 19643357
- [Result] Sogaard P, Egeblad H, Pedersen AK, Kim WY, Kristensen BO, Hansen PS, Mortensen PT. Sequential versus simultaneous biventricular resynchronization for severe heart failure: evaluation by tissue Doppler imaging. Circulation. 2002 Oct 15;106(16):2078-84. doi: 10.1161/01.cir.0000034512.90874.8e. PMID 12379577
- [Result] Sogaard P, Egeblad H, Kim WY, Jensen HK, Pedersen AK, Kristensen BO, Mortensen PT. Tissue Doppler imaging predicts improved systolic performance and reversed left ventricular remodeling during long-term cardiac resynchronization therapy. J Am Coll Cardiol. 2002 Aug 21;40(4):723-30. doi: 10.1016/s0735-1097(02)02010-7. PMID 12204503
- [Result] Haugaa KH, Marek JJ, Ahmed M, Ryo K, Adelstein EC, Schwartzman D, Saba S, Gorcsan J 3rd. Mechanical dyssynchrony after cardiac resynchronization therapy for severely symptomatic heart failure is associated with risk for ventricular arrhythmias. J Am Soc Echocardiogr. 2014 Aug;27(8):872-9. doi: 10.1016/j.echo.2014.04.001. Epub 2014 May 3. PMID 24798865
- [Result] Papadopoulou E, Kaladaridou A, Mattheou J, Pamboucas C, Hatzidou S, Antoniou A, Toumanidis S. Effect of pacing mode and pacing site on torsional and strain parameters and on coronary flow. J Am Soc Echocardiogr. 2015 Mar;28(3):347-54. doi: 10.1016/j.echo.2014.10.014. Epub 2014 Nov 26. PMID 25456534
- [Result] Abraham WT, Adamson PB, Bourge RC, Aaron MF, Costanzo MR, Stevenson LW, Strickland W, Neelagaru S, Raval N, Krueger S, Weiner S, Shavelle D, Jeffries B, Yadav JS; CHAMPION Trial Study Group. Wireless pulmonary artery haemodynamic monitoring in chronic heart failure: a randomised controlled trial. Lancet. 2011 Feb 19;377(9766):658-66. doi: 10.1016/S0140-6736(11)60101-3. PMID 21315441
- [Result] Pappone C, Augello G, Rosanio S, Vicedomini G, Santinelli V, Romano M, Agricola E, Maggi F, Buchmayr G, Moretti G, Mika Y, Ben-Haim SA, Wolzt M, Stix G, Schmidinger H. First human chronic experience with cardiac contractility modulation by nonexcitatory electrical currents for treating systolic heart failure: mid-term safety and efficacy results from a multicenter study. J Cardiovasc Electrophysiol. 2004 Apr;15(4):418-27. doi: 10.1046/j.1540-8167.2004.03580.x. PMID 15089990